CLINICAL TRIAL: NCT05292794
Title: A Multi-Center, Controlled Study to Evaluate Use of CereGate Therapy to Reduce Freezing of Gait in Participants Diagnosed With Parkinson's Disease
Brief Title: Use of CereGate Therapy for Freezing of Gait in PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CereGate Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-001
Record Dates: First submitted 2022-02-23; First posted 2022-03-23 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-10

CONDITIONS: Parkinson Disease; Freezing of Gait; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- PD Patients treated with CereGate Software (Experimental): This singular arm contains participants diagnosed with Parkinson's Disease (PD) and previously implanted with a subthalamic nucleus deep brain stimulation (STN-DBS) System. Participants will use the CereGate software for 60(+/-8) days on demand.
  Interventions: Device: CereGate Software; BSN cDBS Programmer; BSN Burst Programmer

INTERVENTIONS:
Device: CereGate Software; BSN cDBS Programmer; BSN Burst Programmer — CereGate's objective is to, with a single DBS system implanted in the standard STN location for PD:
  (i) deliver conventional tonic DBS stimulation of STN-to mitigate dopamine-responsive symptoms; and concurrently (ii) deliver bursting DBS-induced "cueing" stimulation-to mitigate FOG.
  The sole function of CereGate Software is to guide the clinician through a systematic investigation of the stimulation parameter space to thereby configure / tune CereGate Therapy for each participant. CereGate Software proposes parameters for the clinician to evaluate and assists in documenting the response. It does not send commands to, nor control the output of, the DBS System.

SUMMARY:
A Multi-Center, Controlled Study to Evaluate Use of CereGate Therapy to Reduce Freezing of Gait in Participants Diagnosed with Parkinson's Disease.

DETAILED DESCRIPTION:
This is a multi-center, controlled, study in which participants diagnosed with Parkinson's Disease (PD) and previously implanted with a subthalamic nucleus deep brain stimulation (STN-DBS) System will be assessed prior to initiation of CereGate (CG) therapy, and during CereGate therapy. No randomization will occur in this study.

Participants will complete a total of five study visits (2 Screening Visits, Initiation Visit, day 60 follow-up and day 61 follow-up). The expected duration of participation in the clinical study is up to 104 days for each subject.

Up to 41 participants diagnosed with PD previously implanted with a compatible STN-DBS System will be enrolled at up to eight (8) sites in the United States. A maximum of 15 subjects may be enrolled at any site.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has an implanted STN-DBS system with Boston Scientific Gevia™ or Genus™ R16 IPG connected to any brand lead or extension that have been approved by the FDA to be used with Gevia or Genus IPGs.
2. Participant is receiving treatment with carbidopa/levodopa, and/or with a dopamine agonist at the optimal doses as determined by a movement disorders neurologist.
3. DBS optimized with documented improvement in motor signs (UPDRSIII) from DBS

Exclusion Criteria:

1. Participant is unable to understand the study requirements and the treatment procedures, or unwilling / unable to provide written informed consent before any study-specific tests or procedures are performed.
2. Participant is unwilling or unable to comply with visit schedule and study related procedures.
3. Participant's medication regimen has not been stable for at least 28 days prior to CG initiation.
4. Participant's DBS stimulation settings have not been stable for at least 28 days prior to CG initiation.
5. Participant is less than 21 years of age or older than 80 years of age.
6. Participant is a female who is breastfeeding or of child-bearing potential with a positive urine pregnancy test or not using adequate contraception as determined by the study investigator.
7. Participant has a terminal illness with life expectancy of < 1 year.
8. Participant has history of recurrent or unprovoked seizures.
9. Participant currently diagnosed with drug or alcohol abuse, per DSM-5 criteria.
10. Participant is in a very advanced stage of Parkinson's disease defined as: (i) Stage 5 as classified by the Hoehn and Yahr scale on medication and DBS (non-ambulatory) or (ii) participant requires an assistive device to perform the TBC OFF-meds /ON-DBS at the time of enrollment.
11. Participant has a condition that makes walking difficult or could interfere with the study procedures or confound the evaluation of the study data, including musculoskeletal issues, peripheral neuropathies, hip/knee prostheses, or any visual or anatomical abnormality that affects their walking.
12. Participant has disabling dyskinesias.
13. Participant has a history of suicide attempt or current active suicidal ideation as determined by a positive response to Items 2-5 of suicide ideation sub-scale of the Columbia Suicide Severity Rating Scale (CSSRS).
14. Participant, at the time of enrollment, fails the subthalamic nucleus (STN) stimulation challenge test (subject must perceive distinct bilateral sensations).
15. Participant has less than 8% arrhythmicity as measured in the Turning and Barrier Course Figures of 8 (TBC-F8) pre-CG therapy (ON Medications/ON DBS /OFF CG).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Objective | Pre-CG therapy to post-CG-therapy follow-up Day 60 Visit (Day 60 ± 8)
  The primary objective of this study is to determine whether adjunctive use of CereGate therapy reduces Freezing of Gait in participants diagnosed with Parkinson's Disease in the ON-MEDS/ON-DBS state. The primary efficacy endpoint for this study is the mean percent change in excess arrhythmicity during Turning and Barriers Course Figures of 8 (TBC-F8) while ON-med/ON-DBS, pre-CG therapy to post-CG Therapy follow-up. The Opal wearable inertial measurement sensor (APDM Inc., Portland, OR) will be used to capture kinemetric data, from which the arrhythmicity will be extracted. Excess arrhythmicity will be calculated by subtracting the "normal" arrhythmicity (during TBC-F8 in age-matched controls).

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint | Pre-CG therapy to post-CG-therapy follow-up Day 61 Visit (Day60 Visit +1-8d).
  The secondary objective of this study is to determine whether adjunctive use of CereGate therapy reduces FOG in participants diagnosed with PD as measured by mean percent change in excess arrhythmicity in the OFF-med/ON-DBS state.

OTHER OUTCOMES:
Safety Endpoints | From 1st Screening Visit through Day 61 (Day 60 Visit +1-8d) follow-up visit.
  Safety endpoints for this study will include the following by interventional condition (i.e., CereGate therapy ON or OFF): Proportion of participants who experience one or more stimulation-related serious adverse events (SAEs) Proportion of participants who experience any stimulation related adverse event Proportion of participants who experience each unique type of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Brian Blischak, Study Chair — CereGate Inc.
Locations (7):
- United States (7):
  - Kaiser Permanente, KPNC Comprehensive Movement Disorders Program, Redwood City, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Wake Forest University, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No